CLINICAL TRIAL: NCT07298382
Title: See the Impact Beem's Blue Light Therapy Has on Your Skin Health!
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 46140
Record Dates: First submitted 2025-12-05; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Skin
MeSH Terms: interventions — Phototherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm longitudinal where participants act as their own control (Experimental): Single Arm longitudinal where participants act as their own control
  Interventions: Device: Blue Light Therapy

INTERVENTIONS:
Device: Blue Light Therapy — Blue Light Therapy therapy, combining blue, red, and infrared light, has been backed by studies showing improved skin health and reduced signs of aging. The medical community generally supports light therapy for its non-invasive nature and potential benefits, though results can vary. Social media buzz highlights glowing testimonials, while the general population views it as a promising skincare enhancement with minimal risks. Benefits include improved complexion and reduced acne, with risks being rare and minor, such as temporary redness.
  Treatment:
  First 5 Minutes 450nm (Blue) Second 5 Minutes 450nm (Blue) 660nm (Red) 810nm (Infrared) Final 10 Minutes 660nm (Red) 810nm (Infrared)

SUMMARY:
Participants will experience a rejuvenating twice-weekly light therapy journey that blends the power of blue, red, and infrared light. Each 20-minute session flows through three phases: starting with refreshing blue light to awaken and energize, then moving into soothing red light, and finishing with deeply nourishing infrared light. This unique protocol is designed to help unlock healthier-looking skin and boost your natural glow.

DETAILED DESCRIPTION:
Treatment activities:

Twice a week, for 20 minutes, participants will undergo exposure to blue, red, and infrared light as part of the light therapy treatment.

Assesments and frequency:

Comprehensive Weekly Skin Health Self-Assessment: Conducted weekly. Dermatology Life Quality Index (DLQI): Conducted during the study. Facial Skin Self-Assessment Survey: Conducted during the study. Pre/Post Photos of Participants' Skin: Conducted at the beginning and end of the study.

Methodology:

The study entitled "See the Impact Beem's Blue Light Therapy Has on Your Skin Health!" aims to evaluate the effectiveness of a light therapy regimen on improving skin health. This single-arm observational trial, conducted under Efforia's Signal Phase study design, involves participants undergoing a twice-weekly, 20-minute light therapy session. Each session is structured into three phases: starting with blue light, transitioning to red light, and concluding with infrared light, each targeting different aspects of skin health. By allowing participants to act as their own control, the trial will provide initial insights into the potential benefits of this therapy for enhancing skin appearance and health, with a focus on gathering preliminary efficacy and safety data.

The study's methodology is designed to assess how these light therapies influence skin conditions through a series of personalized assessments and feedback mechanisms. Participants will engage in various self-assessment tasks, including a Comprehensive Weekly Skin Health Self-Assessment, Dermatology Life Quality Index (DLQI) surveys, and Facial Skin Self-Assessment Surveys. These tasks are complemented by pre- and post-therapy photographic documentation to visually track skin changes. By collecting this data, the trial seeks to discern patterns and indications of improvement in skin health, potentially providing a directional indication of positive results from the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Exclusion Criteria:

* Individuals with Epilepsy
* Individuals with Photosensitivity
* Individuals with eye conditions
* Pregnant individuals
* Individuals with skin sensitivity
* Individuals taking certain light-sensitive medications

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-10-06 (Estimated); Study Completion 2026-10-06 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Weekly Skin Health Self-Assessment | Baseline through Day 30 (weekly assessments)
  The Comprehensive Weekly Skin Health Self-Assessment is designed to meticulously evaluate various aspects of skin health, including clarity, breakouts, pore size, redness, moisture, sensitivity, and signs of aging. This detailed survey allows individuals to track changes weekly, providing insights into the effectiveness of their skincare routines and the impact of lifestyle choices on their skin's condition. By regularly monitoring a wide range of skin health indicators, users can make informed adjustments to their skincare practices, aiming for optimal skin health. The survey fosters a proactive approach to skincare, emphasizing the importance of observation and adjustment based on personal skin behavior.
  Scoring scale 0-75 Interpretation Higher score is associated with better perceived skin health Lower score is associated with worse perceived skin health
Dermatology Life Quality Index (DLQI) | Baseline through Day 30 (weekly assessments)
  The Dermatology Life Quality Index (DLQI) is a survey designed to measure the impact of skin-related issues on the quality of life over the past week. It assesses various dimensions of daily living, from personal discomfort to social interactions, influenced by skin conditions. This index is valuable for both patients and healthcare providers to understand the severity and emotional toll of dermatological issues. By quantifying the effects on daily activities and personal relationships, the DLQI helps in guiding treatment decisions and measuring treatment outcomes.
  Scoring Range
  Minimum score: 0
  Maximum score: 30
  Each of the 10 items is scored from 0 to 3, yielding a total score between 0 and 30.
  Score Interpretation
  Higher scores indicate worse outcomes, meaning a greater negative impact of skin disease on a participant's quality of life.
Facial Skin Self-Assessment Survey | Baseline through day 30 (weekly assessments)
  The Comprehensive Weekly Skin Health Self-Assessment is designed to meticulously evaluate various aspects of skin health, including clarity, breakouts, pore size, redness, moisture, sensitivity, and signs of aging. This detailed survey allows individuals to track changes weekly, providing insights into the effectiveness of their skincare routines and the impact of lifestyle choices on their skin's condition. By regularly monitoring a wide range of skin health indicators, users can make informed adjustments to their skincare practices, aiming for optimal skin health. The survey fosters a proactive approach to skincare, emphasizing the importance of observation and adjustment based on personal skin behavior.
  Scoring scale 0-75 Interpretation Higher score is associated with better perceived skin health Lower score is associated with worse perceived skin health

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States